CLINICAL TRIAL: NCT04403256
Title: Changes of Bone-biomarker According to the Severity of Spinal Cord Injury.
Brief Title: Bone-biomarkers of Spinal Cord Injury Patients
Status: Completed | Type: Observational
Sponsor: Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, Dong Gyu Lee, Assistant professor, Yeungnam University Hospital
Other Study IDs: 2019-11-054-001
Record Dates: First submitted 2020-03-25; First posted 2020-05-27 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Spinal Cord Injuries; Bone Resorption; Osteoporosis
Keywords: Sclerostin; osteoporosis; Spinal cord injury; Unloading
MeSH Terms: conditions — Spinal Cord Injuries; Bone Resorption; Osteoporosis; Sclerosteosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with spinal cord injury have a high prevalence of osteoporosis due to chronic skeletal unloading. Recently, various treatment drugs for osteoporosis have been developed. In particular, romosozumab, a sclerostin inhibitor, has been reported to have a high therapeutic effect as an inhibitor of bone resorption while promoting bone formation. However, there are a few research concerning sclerostin of spinal cord injuries patients. Therefore we want to analyze the change of sclerostin as well as factors indicating bone formation and absorption marker in spinal cord injury patient.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury patients
* Functional ambulatory category index of 3 or less

Exclusion Criteria:

* history of using bone absorption medication within the effective period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spinal cord injury difficult to walk
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Serum sclerostin level | 1 year
  Serum sclerostin level in spinal cord injury patients

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided